CLINICAL TRIAL: NCT02600065
Title: Analysis of CMV Infections in Patients Suffering From Brain Tumors and Brain Metastases During and After Radio(Chemo)Therapy
Brief Title: Analysis of CMV Infections in Patients With Brain Tumors or Brain Metastases During and After Radio(Chemo)Therapy
Acronym: GLIO-CMV-01
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: GLIO-CMV-01
Record Dates: First submitted 2015-10-23; First posted 2015-11-09 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2021-04

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Blood Specimen Collection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood for CMV status analysis blood for immunophenotyping serum plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study cohort: All patients who are suffering from brain tumor of brain metastases and are willing to participate.
  The treatment-plan of the underlying disease remained unchanged. Blood draw and MRI from patients at several time points during and after radio(chemo)therapy.
  Interventions: Other: Blood draw and MRI

INTERVENTIONS:
Other: Blood draw and MRI — The study is observational. The treatment-plan of the underlying disease remained unchanged. Blood draw and MRI from patients at several time points during and after radio(chemo)therapy.

SUMMARY:
Radio(chemo)therapy is the standard therapy for both, brain tumors and brain metastases. Neurological decline is observed in these patients and tumor progression or radiotherapy side effects have been made responsible for this. However CMV encephalitis may also be a reason. Therefore the investigators aim to analyze the CMV status in patients during and after radio(chemo)therapy. It will be checked by CMV-DNA (PCR analysis) and CMV antibodies (IgG and IgM ELISA) in the blood of the patients. These findings will be correlated with changes in the brain, visualized by MRI. In addition a detailed immunophenotyping in the peripheral blood will be performed.

ELIGIBILITY:
Inclusion Criteria:

* brain tumours (glioblastoma or anaplastic astrocytoma)
* brain metastases from diagnosed primary tumours
* legal age
* planned chemoradiation and adjuvant chemotherapy [metastases]
* planned chemoradiation and adjuvant chemotherapy with temodal (according to Stupp et. al.) [brain tumors]

Exclusion Criteria:

* fertile patients who refuse effective contraception during study treatment
* persistent drug and/or alcohol abuse
* patients not able or willing to behave according to study protocol
* patients in care
* patients that are not able to speak German
* patients with claustrophobia
* patients with artificial joint or any metal parts in the body
* patients with pacemakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain tumours (glioblastoma or anaplastic astrocytoma Patients with brain metastases from diagnosed primary tumours
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2014-11; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of CMV status during radio(chemo)therapy (RCT) | up to day 45 after start of Radiotherapy
  CMV infection will be monitored by virus analysis by an approved laboratory. The analyses were conducted at time points during and after RCT - before RT (day 0), during RT (dose halftime), end of RT (last day of RT), month 3 and 6 after completed RT. This scheme is repeated if patient receives additional RT for relapse treatment. The time points during RT were determined depending on the applied irradiation dose. For glioblastoma the halftime of RT is usually day 23 (received dose 30 Gy) and the end of therapy is usually day 45 (received dose 60 Gy). For cerebral metastases the halftime of the RT is usually day 8 (received dose 9 Gy) and day 16 at the end of therapy (received dose 18 Gy). However, the time points are strongly connected to the received dose.

SECONDARY OUTCOMES:
Change of circulating immune cells of treated patients by deep immunophenotyping. | up to month 6 after the start of Radiotherapy
  Immunophenotyping of the patients. Detection of about 30 distinct immune sell (sub)types together with their activation markers.The analyses were conducted at time points during and after RCT - before RT (day 0), during RT (dose halftime), end of RT (last day of RT), month 3 and 6 after completed RT. This scheme is repeated if patient receives additional RT for relapse treatment. The time points during RT were determined depending on the applied irradiation dose. For glioblastoma the halftime of RT is usually day 23 (received dose 30 Gy) and the end of therapy is usually day 45 (received dose 60 Gy). For cerebral metastases the halftime of the RT is usually day 8 (received dose 9 Gy) and day 16 at the end of therapy (received dose 18 Gy). However, the time points are strongly connected to the received dose.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Prof., Principal Investigator — Department of Radiation Oncology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Departement of Radiation Oncology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided